CLINICAL TRIAL: NCT02474459
Title: Mobile Decision Support System for Nurse Management of Neuromodulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Florida (Other); National Institute of Nursing Research (NINR) (NIH); Wake Forest University Health Sciences (Other); Baylor College of Medicine (Other); NYU (Unknown); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Christopher Butson, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 82859; R01NR014852 (NIH); NCT02066779 (obsolete NCT alias)
Record Dates: First submitted 2015-06-14; First posted 2015-06-17 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; DBS; STN; GPi; Globus pallidus; Subthalamic nucleus; Neuromodulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iPad-based Clinical Support Care (Active Comparator): Subjects in this treatment arm will receive deep brain stimulation (DBS) programming at regular intervals as part of routine clinical care. DBS stimulation programming will be performed using an iPad-based decision support system. Outcomes will be measured using the Unified Parkinson's Disease Rating Scale (UPDRS), Parkinson's Disease Questionnaire (PDQ-39) and the Multi-Dimensional Caregiver Strain Index (MCSI).
  Interventions: Device: iPad-Based Clinical Support Care
- Standard Clinical Care (Active Comparator): Subjects in this treatment arm will receive DBS programming at regular intervals as part of routine clinical care. Outcomes will be measured using the Unified Parkinson's Disease Rating Scale (UPDRS), Parkinson's Disease Questionnaire (PDQ-39) and the Multi-Dimensional Caregiver Strain Index (MCSI).
  Interventions: Other: Standard Clinical Care

INTERVENTIONS:
Device: iPad-Based Clinical Support Care — Subjects in this treatment arm will receive deep brain stimulation (DBS) programming at regular intervals as part of routine clinical care. DBS stimulation programming will be done with the use of a iPad-based decision support system.
  Other Names: iPad-Based Tool
  Arms: iPad-based Clinical Support Care
Other: Standard Clinical Care — Subjects in this treatment arm will receive DBS programming at regular intervals as part of routine clinical care.
  Arms: Standard Clinical Care

SUMMARY:
The purpose of this study is to test the use of a clinical decision support tool for postoperative care of Parkinson's disease patients who are treated using deep brain stimulation (DBS). The central hypothesis is that the use of a DBS clinical decision support system for individual patient management will enable considerable time savings and reduced burden on patients and caregivers.

DETAILED DESCRIPTION:
The proposed study will evaluate outcomes for Parkinson's disease (PD) patients who are treated with unilateral deep brain stimulation (DBS); patients who consent to the study will be randomized to standard care or the experimental group. The study will occur in two phases.

Phase I:

Both the standard care and experimental groups will be medically evaluated identically, but the programming will be different between the groups as the experimental group will be programmed using the iPad. Patients in the control and experimental groups will be monitored with the same frequency at each participating clinic. Data and safety monitoring is the responsibility of each participating PI and the lead PI as the protocol involves minimal risk or no more than a minor increase over minimal risk. We anticipate that a single nurse at each site will perform DBS programming.

Phase II:

Patients in the experimental group will be evaluated and programmed by home health nurses in the patient's home setting. Neurological exams in the clinic will be performed at the first post-operative DBS programming session and 6 months later (the proposed end of the experimental period for each patient). During the intervening period, DBS programming and patient evaluations will be performed by a home health nurse. during this phase, data and safety monitoring will be conducted by a DSMB, which will meet regularly to review all cases and ensure safety. All subjects will be recruited directly through the participating sites' clinic systems, and all subjects will have oral and written informed consent before participation in the study. We anticipate that up to two home health registered nurses (RNs) will be performing DBS programming in phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Planning to receive a DBS device at a participating site.
* Had a DBS device implanted, at a participating site, that hasn't been programmed yet

Exclusion Criteria:

* Had a DBS device implanted at a non-participating site.
* Any previous DBS programming

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Phase I: Difference in deep brain stimulation (DBS) programming time. | 6 months
  Phase I: Difference in deep brain stimulation (DBS) programming time compared to standard care when the DBS programming nurse uses an iPad based decision support system.
Phase II: Difference in number of times the patient travels to the clinic. | 6 months
  Phase II: Difference in total number of times the patient travels to the University of Florida Movement Disorders clinic during the six month study period, except at baseline and 6 months (which were in clinic for everyone).

SECONDARY OUTCOMES:
Differences in caregiver strain for DBS patients using the iPad-based clinical decision support tool | 6 months
  The Multi-Dimensional Caregiver Strain Index (MCSI) is an 18-question self-report scale with 6 subscales of caregiver strain: physical strain, social constraints, financial strain, time constraints, interpersonal strain, and elder demanding/manipulative behavior. A higher score is considered indicative of a greater caregiver strain. MCSI scores range from 0 to 72. Higher scores indicate worse outcomes.
Differences in outcomes for patients in the intervention groups compared to standard care as measured using the Unified Parkinson's Disease Rating Scale (UPDRS) | 6 months
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a rating scale used to follow the longitudinal course of Parkinson's disease. The UPDRS is made up of 5 sections: (1) Evaluation of Mentation, behavior, and mood; (2) Self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, cutting food; (3) Clinician-scored monitored motor evaluation; (4) Hoehn and Yahr staging of severity of Parkinson disease; (5) Schwab and England ADL scale. The higher the UPDRS score, the greater the disability from PD. UPDRS scores range from 0 to 199. Higher scores indicate worse outcomes.
Differences in patient quality of life as measured by the Parkinson's Disease Questionnaire - 39 (PDQ-39). | 6 months
  The Parkinson's Disease Questionnaire - 39 (PDQ-39) is a patient self-reported rating scale that measures impairment in quality of life caused by Parkinson's disease. Scores range from 0 to 100. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Butson, PhD, Principal Investigator — University of Utah Scientific Computing and Imaging Institute
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - University of Florida Center for Movement Disorders & Neurorestoration, Gainesville, Florida
  - NYU Langone Medical Center, New York, New York
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Imaging and Neurosciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duffley G, Lutz BJ, Szabo A, Wright A, Hess CW, Ramirez-Zamora A, Zeilman P, Chiu S, Foote KD, Okun MS, Butson CR. Home Health Management of Parkinson Disease Deep Brain Stimulation: A Randomized Clinical Trial. JAMA Neurol. 2021 Aug 1;78(8):972-981. doi: 10.1001/jamaneurol.2021.1910. PMID 34180949